CLINICAL TRIAL: NCT06339281
Title: A Multicenter Clinical Study of Apatinib Mesylate in Combination With a Physician's Choice Regimen for Her-2 Negative, HR-positive Progressive Breast Cancer.
Brief Title: A Multicenter Clinical Study of Apatinib Mesylate Combined With Doctor's Choice for Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Huiping (Other)
Responsible Party: Sponsor-Investigator, Li Huiping, Director of breast oncology department, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023YJZ87
Record Dates: First submitted 2024-03-05; First posted 2024-04-01 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Breast Cancer
Keywords: Her-2 negative, HR positive , advanced breast cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib mesylate combined with chemotherapy (Capecitabine/vinorelbine) (Experimental)
  Interventions: Drug: apatinib mesylate+Capecitabine Tablets
- Apatinib mesylate combined with endocrine (Active Comparator)
  Interventions: Drug: apatinib mesylate+Fulvestrant injection

INTERVENTIONS:
Drug: apatinib mesylate+Capecitabine Tablets — Apatinib Mesylate Tablets: 500 mg, qd, orally until disease progression or intolerable adverse reactions.
  Capecitabine Tablets: 1000 mg/m2, po, twice a day, d1-d14, discontinued for 1 week after 2 weeks of treatment;
  Arms: Apatinib mesylate combined with chemotherapy (Capecitabine/vinorelbine)
Drug: apatinib mesylate+Fulvestrant injection — Apatinib Mesylate Tablets: 500 mg, qd, orally until disease progression or intolerable adverse reactions.
  Fulvestrant injection 500 mg, intramuscular injection, q4w, once on d1 and d15 in the first cycle;
  Arms: Apatinib mesylate combined with endocrine

SUMMARY:
Previous studies have found good efficacy of (investigator's choice of chemotherapy, or endocrine drug) in combination with apatinib mesylate in the treatment of her-2 negative, chest wall metastatic advanced breast cancer, and the present study proposes to further explore the efficacy of apatinib mesylate in her-2 negative, HR-positive advanced breast cancer.

DETAILED DESCRIPTION:
In order to further explore the efficacy of apatinib mesylate in advanced breast cancer with negative her-2 and positive HR, this study intends to carry out an observation study on the efficacy of apatinib mesylate combined with doctor's choice scheme in the treatment of advanced breast cancer with negative her-2 and positive HR.

ELIGIBILITY:
Inclusion Criteria：

1. Histologically or cytologically confirmed her-2 negative, HR-positive progressive breast cancer (prior chemotherapy (including adjuvant or neoadjuvant) with anthracycline and/or paclitaxel required);
2. No more than 3 lines of chemotherapy for recurrent or metastatic breast cancer;
3. Must have progression previously used endocrine therapy and CDK4/6 inhibitors for recurrent or metastatic disease ;
4. PET-CT（SUV）>5;
5. Age ≥18 years;
6. ECOG PS 0-1;
7. life expectancy ≥ 3 months
8. Have at least one measurable lesion as a target lesion confirmed by CT or MRI according to RECIST version 1.1 criteria. If the target lesion is a lymph node require a short diameter greater than 1.5 ，and the target lesion is not amenable to surgical treatment; the target lesion has not received radiotherapy or has recurred in the radiotherapy field;
9. Appropriate hematopoiesis；
10. Appropriate liver function；
11. Appropriate renal function；
12. Normal coagulation;
13. Females of childbearing potential willing to use contraception during the trial: negative serum or urine pregnancy test within 7 days prior to dosing.

Exclusion Criteria:

1. Received radiation therapy within 28 days prior to enrollment. Radiotherapy for the relief of metastatic bone pain prior to enrollment is permitted, provided that no more than 30% of the total marrow-containing bone is irradiated, with the exception of patients with good bone feel prior to treatment;
2. The presence of evidence of central nervous system metastases;
3. Current or recent (within 30 days prior to enrollment) use of another investigational drug or participation in another clinical study
4. Other malignancy within 5 years (except adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or controlled basal cell carcinoma of the skin)
5. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg despite optimal pharmacologic therapy)
6. Myocardial ischemia or myocardial infarction of class II or greater, poorly controlled arrhythmias (including qtc intervals ≥450 ms in men and ≥470 ms in women);
7. Grade III-IV cardiac insufficiency according to NYHA criteria, or cardiac ultrasound suggesting left ventricular ejection fraction (LVEF) <50%;
8. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or under thrombolytic or anticoagulant therapy;
9. Have had clinically significant bleeding symptoms or a definite bleeding tendency within the previous 3 months, such as gastrointestinal bleeding, bleeding gastric ulcer, fecal occult blood +++ or more at baseline, or have vasculitis
10. Have undergone major surgical procedures or have sustained a severe traumatic injury, fracture, or ulcer within the previous 4 weeks
11. Having factors that significantly affect the absorption of oral medication, such as inability to swallow, chronic diarrhea and intestinal obstruction, etc;
12. Urine routine suggestive of urinary protein ≥ ++, or confirmed 24-hour urine protein volume ≥ 1.0 g;
13. Plasmapheresis (including pleural fluid, ascites, and pericardial effusion) that is clinically symptomatic and requires surgical management;
14. Other conditions that, in the judgment of the investigator, may affect the conduct of the clinical study and the determination of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 36 months
  Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, MD, Study Chair — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: No
The research plan will be shared after the patient registration is completed.